CLINICAL TRIAL: NCT06049615
Title: The Conscious Sedation Single Arm Sub-Study
Brief Title: Conscious Sedation Study
Acronym: CSS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Conformal Medical, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C-006
Record Dates: First submitted 2023-07-29; First posted 2023-09-22 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: The Conscious Sedation Single Arm Sub-Study is designed to evaluate the safety and performance of the CLAAS device implantation procedure using conscious sedation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- CLAAS (Experimental): Subjects to be implanted with the CLAAS device.
  Interventions: Device: CLAAS® System

INTERVENTIONS:
Device: CLAAS® System — The CLAAS® System delivers a plug to the ostia of the Left Atrial Appendage (LAA) and is designed to occlude the appendage to eliminate blood flow. It is designed to conform to the geometry of the LAA. The implant is designed to permanently seal off the LAA from the LA with an endothelial layer that forms across the LA face of the implant. The implant is available in two different sizes; Regular (27mm) and Large (35mm) to accommodate patient anatomy. Angiography and/or echocardiography may be used to determine the LAA ostium diameter to properly select the Implant size. The implant has an inner, cylindrical, Nitinol endoskeleton that provides the mechanical base structure. The Nitinol endoskeleton contains 10 face struts and 20 anchors (Regular) and 12 struts and 24 anchors (Large) facing proximally to engage the tissue to resist movement. The endoskeleton also provides the conformable structure to enable the foam cylinder to compress against the LAA tissue to facilitate sealing.

SUMMARY:
The Conscious Sedation Single Arm Sub-Study is designed to evaluate the safety and performance of the CLAAS device implantation procedure using conscious sedation.

DETAILED DESCRIPTION:
The Sub-Study is a prospective single arm trial evaluating a conscious sedation protocol. The Sub-Study will evaluate the safety and performance of the CLAAS device using conscious sedation in comparison with the device delivery safety and performance observed in the CLAAS arm of the RCT. The Sub-Study will be performed in accordance with all protocol requirements and all subjects will be evaluated for Primary Endpoint based on the product performance at the 45 days post procedure assessment. Enrollment in the Sub-Study will not commence until enrollment in the randomized cohort is complete, initial safety of the CLAAS system is confirmed by the DSMB and FDA approval of the Sub-Study has been granted through an IDE Supplement. All subjects enrolled in the conscious sedation single arm study will follow the same clinical protocol requirements and follow-up as the randomized subjects. The Sub-Study will be identified by an NCT that is separate from the RCT with Roll-in.

ELIGIBILITY:
General Inclusion Criteria

1. Male or non-pregnant female aged ≥18 years.
2. Documented non-valvular AF (paroxysmal, persistent, or permanent).
3. High risk of stroke or systemic embolism, defined as CHADS2 score of ≥2 or CHA2DS2-VASc score of ≥3.
4. Has an appropriate rationale to seek a non-pharmacologic alternative to long-term oral anticoagulation.
5. Deemed by the site investigator to be suitable for short term oral anticoagulation therapy but deemed less favorable for long-term oral anticoagulation therapy .
6. Deemed appropriate for LAA closure by the site investigator and a clinician not a part of the procedural team using a shared decision-making process in accordance with standard of care.
7. Able to comply with the protocol-specified medication regimen and follow-up evaluations.
8. The patient (or legally authorized representative, where allowed) has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent approved by the appropriate Institutional Review Board (IRB)/Regional Ethics Board (REB).

General Exclusion Criteria

1. Pregnant or nursing patients and those who plan pregnancy in the period up to one year following the index procedure. Female patients of childbearing potential must have a negative pregnancy test (per site standard test) within 7 days prior to index procedure.
2. Anatomic conditions that would prevent performance of an LAA occlusion procedure (e.g., prior atrial septal defect [ASD] or high-risk patent foramen ovale [PFO] surgical repair or implanted closure device, or obliterated or ligated left atrial appendage).
3. Atrial fibrillation that is defined by a single occurrence or that is transient or reversible (e.g., secondary thyroid disorders, acute alcohol intoxication, trauma, recent major surgical procedures).
4. A medical condition (other than atrial fibrillation) that mandates long-term oral anticoagulation (e.g., history of unprovoked deep vein thrombosis or pulmonary embolism, or mechanical heart valve).
5. History of bleeding diathesis or coagulopathy, or patients in whom antiplatelet and/or anticoagulant therapy is contraindicated.
6. Documented active systemic infection.
7. Symptomatic carotid artery disease (defined as >50% stenosis with symptoms of ipsilateral transient or visual TIA evidenced by amaurosis fugax, ipsilateral hemispheric TIAs or ipsilateral stroke); if subject has a history of carotid stent or endarterectomy the subject is eligible if there is <50% stenosis noted at the site of prior treatment.
8. Recent (within 30 days of index procedure) or planned (within 60 days post-procedure) cardiac or major non-cardiac interventional or surgical procedure.
9. Recent (within 30 days of index procedure) stroke or transient ischemic attack.
10. Recent (within 30 days of index procedure) myocardial infarction.
11. Vascular access precluding delivery of implant with catheter-based system.
12. Severe heart failure (New York Heart Association Class IV).
13. Prior cardiac transplant, history of mitral valve replacement or transcatheter mitral valve intervention, or any mechanical valve implant.
14. Renal insufficiency, defined as estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2 (by the Modification of Diet in Renal Disease equation).
15. Platelet count <75,000 cells/mm3 or >700,000 cells/mm3, or white blood cell count <3,000 cells/mm3.
16. Known allergy, hypersensitivity or contraindication to aspirin, heparin, or device materials (e.g., nickel, titanium) that would preclude any P2Y12 inhibitor therapy, or the patient has contrast sensitivity that cannot be adequately pre-medicated.
17. Actively enrolled or plans to enroll in a concurrent clinical study in which the active treatment arm may confound the results of this trial.
18. Unable to undergo general anesthesia.
19. Known other medical illness or known history of substance abuse that may cause non-compliance with the protocol or protocol-specified medication regimen, confound the data interpretation, or is associated with a life expectancy of less than 5 years.
20. A condition which precludes adequate transesophageal echocardiographic (TEE) assessment.

Echocardiographic Exclusion Criteria

1. Left atrial appendage anatomy which cannot accommodate a commercially available control device or the CLAAS device per manufacturer IFU (e.g., the anatomy and sizing must be appropriate for both devices to be enrolled in the trial).
2. Intracardiac thrombus or dense spontaneous echo contrast consistent with thrombus, as visualized by TEE prior to implant.
3. Left ventricular ejection fraction (LVEF) <30%.
4. Moderate or large circumferential pericardial effusion >10 mm or symptomatic pericardial effusion, signs or symptoms of acute or chronic pericarditis, or evidence of tamponade physiology
5. Atrial septal defect that warrants closure.
6. High risk patent foramen ovale (PFO), defined as an atrial septal aneurysm (excursion >15 mm or length >15 mm) or large shunt (early [within 3 beats] and/or substantial passage of bubbles, e.g., ≥20).
7. Moderate or severe mitral valve stenosis (mitral valve area <1.5cm2).
8. Complex atheroma with mobile plaque of the descending aorta and/or aortic arch.
9. Evidence of cardiac tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy: Evaluating the Performance of CLAAS, as defined below: | 7 days through 45 days post-procedure
  1. Successful implantation of the LAAO Device in the LAA with acceptable position (e.g. as measured at LAA orifice) through 45 days post-procedure
  2. Complete closure or peri-device residual leak ≤5 mm in width on TEE, as evaluated by independent core lab at 45 days post-procedure
  3. Without in-hospital major procedure-related complications during hospitalization or at 7 days, whichever is first
Primary Safety: A Composite of Major Procedure-Related Complications Assessed through 45-Days | 45 days post procedure
  A composite of Major Procedure-related complications assessed through 45 days (listed below) as adjudicated by an independent Clinical Events Committee as related to either the study device or procedure.
  Major Procedure-Related Complications includes any of the following specific events with the specific definitions outlined for each component:
  * cardiac perforation,
  * pericardial effusion requiring drainage,
  * ischemic stroke,
  * device embolization,
  * major vascular complications